CLINICAL TRIAL: NCT05054088
Title: ImmuneSense™ COVID-19 Variant Study
Brief Title: ImmuneSense COVID-19 Variant Study
Status: Completed | Type: Observational
Sponsor: Adaptive Biotechnologies (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-00974
Record Dates: First submitted 2021-09-20; First posted 2021-09-23 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Covid19
Keywords: Variant
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood will be collected in volumes of 5 mL (1 x 10 mL K2 EDTA tube) for each participant. It will be considered a protocol deviation if less than 2mL of whole blood is collected per tube All whole blood samples collected during the study visit will be shipped ambiently to Adaptive. Upon arrival at Adaptive, blood will undergo DNA extraction, and the T-Detect TM COVID test will be performed as applicable and per laboratory protocols. Additional assays may be applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Subjects who have tested positive for SARS-CoV-2 by EUA RT-PCR testing with symptoms compatible with SARS-CoV-2 infection.
  Interventions: Device: T-Detect COVID test
- Cohort 2: Subjects who have tested positive for SARS-CoV-2 by EUA RT-PCR testing with symptoms compatible with SARS-CoV-2 infection.
  Interventions: Device: T-Detect COVID test

INTERVENTIONS:
Device: T-Detect COVID test — • The T-DetectTM COVID test is an EUA granted investigational device that is indicated to assess a T-cell immune response to SARS-CoV-2 via the testing of blood samples from patients with signs and symptoms of suspected COVID-19.

SUMMARY:
This study will assess the clinical performance of the T-Detect™ COVID test to identify an immune response to SARS-CoV-2 infection in the setting of multiple circulating variants of the SARS-CoV-2 virus. Performance may vary depending on the variants circulating at the time of testing, including newly emerging strains of SARS-CoV-2 and their prevalence, which changes over time.

ELIGIBILITY:
General Inclusion Criteria

Inclusion Criteria:

Participants must satisfy the following criteria to be enrolled in the study:

i. Individuals who have tested positive for SARS-CoV-2 via EUA RT-PCR testing. ii. Male and female participants of any race and ethnicity between 18 to 89 years of age (inclusive) at the time of enrollment in the study. iii. Must be able to communicate with the investigator, understand, and comply with the requirements of the study. iv. Must be able to provide estimated date of symptom onset. v. Must be available for specimen collection greater than 14 days (i.e., 15 days inclusive onward) and less than 107 days (i.e., 106 days inclusive or less) after first exhibiting symptoms of confirmed SARS-CoV-2 infection.

Exclusion Criteria:

The presence of any of the following will exclude a participant from enrollment:

* Individuals who did not test positive for SARS-CoV-2 on EUA RT-PCR.
* Protected populations including pregnant women, prisoners, mentally disabled persons, and wards-of-the state.
* Any significant condition, laboratory abnormality, or psychiatric illness that would prevent the participant from safely participating in the study.
* Exposure to a SARS-CoV-2 investigational drug (new chemical entity) within 60 days prior to enrollment at the discretion of the Sponsor.
* Receipt of immunosuppressive medications, such as, but not limited to, recent moderate- or high-dose systemic steroids or immunomodulators within 1 month prior to enrollment at the discretion of the Sponsor.
* Treatment with immunosuppressants/ immunomodulators that do not impact T cells or B cells may be allowed at the discretion of the Sponsor.
* Steroid formulations including low-dose oral steroids (≤ 10 mg prednisone equivalents per day), inhaled steroids, or topical steroids are not considered exclusionary. Doses >10 and <20 mg prednisone equivalents per day, must receive Sponsor approval.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospective ascertainment of a target of 50 whole blood samples (1 sample per individual), and a maximum number of 250 whole blood samples, from individuals between the ages of 18-89 who reside within the United States who have tested positive for SARS-CoV-2 infection via RT-PCR test.
  Pregnant women, prisoners, mentally disabled persons, and wards-of-the-state will be excluded to prevent any risk to these vulnerable populations.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Primary Objective: Positive Percent Agreement | Baseline
  To determine the positive percent agreement (PPA) of the T-Detect™ COVID test with SARS-CoV-2 RT-PCR testing in populations having multiple circulating SARS-CoV-2 variant strains. The primary endpoint is the positive percent agreement (PPA) of the T-Detect™ COVID test with SARS-CoV-2 RT-PCR testing.

CONTACTS AND LOCATIONS:
Overall Officials: Darcy Gill, PhD, Principal Investigator — Adaptive Biotechnologies
Locations (15):
- United States (15):
  - Decentralized Trial Model- Phoenix, Phoenix, Arizona
  - Decentralized Trial Model- Fullerton, Fullerton, California
  - Decentralized Trial Model- California, Los Angeles, California
  - Decentralized Trial Model- Modesto, Modesto, California
  - Decentralized Trial Model- Sacramento, Sacramento, California
  - Decentralized Trial Model- California, San Diego, California
  - Decentralized Trial Model- San Francisco, San Francisco, California
  - Decentralized Trial Model- Denver, Denver, Colorado
  - Decentralized Trial Model - Washington D.C., Washington D.C., District of Columbia
  - Decentralized Trial Model- Florida, Miami, Florida
  - Decentralized Clinical Trial Model- New York City, New York, New York
  - Decentralized Trial Model- Portland, Portland, Oregon
  - Decentralized Trial Model- Utah, Salt Lake City, Utah
  - Decentralized Trial Model- Seattle, Seattle, Washington
  - Decentralized Trial Model- Vancouver, WA, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: No